CLINICAL TRIAL: NCT01615055
Title: Prevention of Cognitive Decline After Chemotherapy, With Fluoxetine Treatment
Brief Title: Fluoxetine Prevention Trial
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study withdrawn. No participants enrolled.
Sponsor: University of California, Los Angeles (Other)
Collaborators: City of Hope Medical Center (Other)
Responsible Party: Principal Investigator, Daniel H. Silverman, Professor, Medical and Molecular Pharmacology, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 12-000568
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Cognitive Dysfunction
Keywords: Chemotherapy; Cognitive; Prozac; Fluoxetine; FDG; PET
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Fluoxetine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Fluoxetine tablets (Experimental)
  Interventions: Drug: Fluoxetine
- Placebo tablets (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Fluoxetine — 20-40 mg fluoxetine po qd for 6 months
  Other Names: Prozac
  Arms: Fluoxetine tablets
Other: Placebo — 20-40 mg pharmacologically inactive tablets for 6 months
  Other Names: "sugar" pill
  Arms: Placebo tablets

SUMMARY:
Many cancer survivors are experiencing problems with memory and other cognitive abilities following cancer treatment. Little is known concerning the contributions of potentially preventive therapies on cognitive function, but animal studies have pointed to the potential value of the medication fluoxetine in this context. We aim to determine whether six months of fluoxetine therapy can preserve brain function in patients who have undergone chemotherapy, and examine potential biological mechanisms for its protective effects in humans. If use of fluoxetine in cancer patients can be validated in this manner, it will represent the first drug demonstrated to prevent cerebral dysfunction associated with exposure to chemotherapy. Moreover, as this involves an agent that is already FDA-cleared for other indications, widely commercially available throughout the U.S. and other parts of the world, and relatively inexpensive since it is obtainable in generic formulations, it would represent a pharmacologic approach that is amenable to rapid translation to the clinical setting.

DETAILED DESCRIPTION:
Systematic studies of adverse cognitive and neurobiological changes subsequent to chemotherapy for lymphoma, breast, and other cancers have attracted substantial interest in the past decade. Little is known, however, concerning the feasibility and effects of potentially protective therapies on cerebral function in patients undergoing chemotherapy. Animal models have recently proved useful in examining some of the toxic effects of chemotherapy agents on working memory and other abilities, as well as on biological properties such as proliferation and survival of neuronal precursors involved in hippocampal neurogenesis. Such models have also proved useful for testing potential neuroprotective properties of agents given before, during and/or after chemotherapy. For example, impairment in spatial working memory and decreased hippocampal neurogenesis is induced in rats by the chemotherapy agent methotrexate, but co-administration of the (FDA-cleared and commercially available) drug fluoxetine has been shown to counteract the negative long-term effects on memory and hippocampal neurogenesis otherwise occurring after methotrexate administration. To determine whether such a strategy could be effective in counteracting effects that chemotherapy may have on cerebral function in humans, well-controlled experimental data obtained with cancer patients is needed.

This investigation will employ a prospective, randomized, double-blinded, placebo-controlled design, to provide a rigorous test of whether fluoxetine, a drug with a long-standing excellent safety profile in humans most commonly marketed as an antidepressant, can offer protection to breast cancer or lymphoma patients against changes in cerebral function occurring after chemotherapy (Specific Aim 1). It will further provide a test of the durability of any protective effects beyond the period during which fluoxetine is used, by re-assessing function approximately 6 months after completion of the regimen (Specific Aim 2). Cerebral function will be assessed by determining distributions of regional cerebral metabolism, previously demonstrated to sensitively detect functional alterations and closely reflect diminished cognitive abilities with high statistical power, using positron emission tomography with the glucose analog radiotracer [F-18]fluorodeoxyglucose. Neuropsychologic testing will be conducted in parallel with neuroimaging studies and, as a step towards understanding mechanisms underlying neurotoxic effects of chemotherapy and potentially related to protective effects of fluoxetine, peripheral markers of inflammatory cytokines will be measured in blood samples drawn at the time of neuroimaging (Specific Aim 3). If use of fluoxetine in cancer patients can be validated in this manner and lead to its adoption in the clinical setting, it will constitute the first drug with demonstrated utility for the prevention of cerebral dysfunction associated with exposure to chemotherapy. Moreover, as this involves an agent that is already FDA-cleared for other indications, widely commercially available throughout the U.S. and other parts of the world, and relatively inexpensive since it is obtainable in generic formulations, it would represent a pharmacologic approach that is amenable to rapid translation to the clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo chemotherapy, or has completed chemotherapy no more than a month prior to enrollment, for breast cancer or lymphoma
* Age 21 or above
* Geographically accessible for follow-up in one year
* English language proficient
* Able to provide informed consent

Exclusion Criteria:

* Pregnant
* Evidence of current or past disorder/disease of the central nervous system or any medical condition that might be expected to impact cognitive functioning (e.g. multiple sclerosis)
* History of head trauma with loss of consciousness greater than 30 minutes
* Epilepsy, dementia, or severe learning disability
* Current psychotic-spectrum disorder (e.g. schizophrenia, bipolar disorder, major affective disorder) or current substance abuse or dependence
* History of whole brain irradiation or surgery
* Active diagnosis of autoimmune disorder e.g., systemic lupus erythematosis, rheumatoid arthritis, vasculitis
* Insulin dependent diabetes
* Uncontrolled allergic condition or asthma
* Chronic use of oral steroid medication
* Hormone therapy (estrogen, progestin compounds) other than vaginal estrogen
* Due to the subtleties of neuropsychological test evaluation, including necessity for repeated administration with alternate forms, we must also exclude non-English language proficient subjects.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in regional cerebral metabolism | Baseline and 6 months

SECONDARY OUTCOMES:
Durability of the protective effect of fluoxetine | 6 months and 1 year
Change from baseline in neuropsychological (cognitive, functional) test results | Baseline, 6 months, and 1 year
Correlation between cognitive functioning and cerebral metabolism by correlating neuropsychological testing results with PET imaging | Baseline, 6 months, and 1 year
Correlation between inflammatory cytokines and cerebral metabolism by correlating blood cytokine marker levels with PET imaging | Baseline, 6 months, and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Daniel H. Silverman, M.D., Ph.D., Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - City of Hope, Duarte, California
  - UCLA Medical Center, Los Angeles, California